CLINICAL TRIAL: NCT01709214
Title: A Randomized, Double-Blind, Placebo- and Active Controlled Study to Evaluate the Safety and Efficacy of GRT6005 in Patients With Moderate to Severe Chronic Pain Due to Osteoarthritis of the Knee
Brief Title: Safety and Efficacy Study of GRT6005 in Patients With Osteoarthritis (OA) Knee Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tris Pharma, Inc. (Industry)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GRT-MD-101
Record Dates: First submitted 2012-10-16; First posted 2012-10-18 (Estimated); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Moderate to Severe Chronic Pain Due to Osteoarthritis of the Knee
Keywords: Osteoarthritis; Knee; Pain; Chronic; OA; Arthritis
MeSH Terms: conditions — Osteoarthritis; Pain; Bronchiolitis Obliterans Syndrome; Arthritis | interventions — 6'-fluoro-4',9'-dihydro-N,N-dimethyl-4-phenylspiro(cyclohexane-1,1'(3'H)-pyrano(3,4-b)indol)-4-amine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cebranopadol (GRT6005) Low-Dose Range (Experimental): Once daily GRT6005, flexible dosing 200, 300 or 400 micrograms, and once daily Placebo; oral administration for 15 weeks
  Interventions: Drug: Cebranopadol (GRT6005) Low-Dose Range; Drug: Placebo
- Cebranopadol (GRT6005) High-Dose Range (Experimental): Once daily GRT6005, flexible dosing 400, 600 or 800 micrograms, and once daily Placebo; oral administration for 15 weeks
  Interventions: Drug: Cebranopadol (GRT6005) High-Dose Range; Drug: Placebo
- Placebo (Placebo Comparator): Twice daily Placebo, oral administration for 15 weeks
  Interventions: Drug: Placebo
- Oxycodone CR (Active Comparator): Twice daily Oxycodone CR, flexible dosing 10, 20, 30, 40 or 50 milligrams; oral administration for 15 weeks
  Interventions: Drug: Oxycodone CR

INTERVENTIONS:
Drug: Cebranopadol (GRT6005) Low-Dose Range — Capsules
  Arms: Cebranopadol (GRT6005) Low-Dose Range
Drug: Cebranopadol (GRT6005) High-Dose Range — Capsules
  Arms: Cebranopadol (GRT6005) High-Dose Range
Drug: Placebo — Capsules that did not contain active substance but appeared identical to the cebranopadol and oxycodone CR capsules
  Arms: Cebranopadol (GRT6005) High-Dose Range; Cebranopadol (GRT6005) Low-Dose Range; Placebo
Drug: Oxycodone CR — Capsules containing oxycodone CR 10 or 20 milligrams
  Arms: Oxycodone CR

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of GRT6005 compared to placebo in patients with moderate to severe chronic pain due to osteoarthritis (OA) of the knee. This study includes a maximum 21 day Screening Period followed by a 15-week Double-blind Treatment Period and a 4-7 day Safety Follow-up period. Patients who are eligible for the Double-blind Treatment Period will be randomized to one of following treatment groups: GRT6005 high-dose range (400, 600 or 800 mcg), GRT6005 low-dose range (200, 300 or 400 mcg), oxycodone controlled release (CR) dose range (10, 20, 30, 40 or 50 mg) or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of osteoarthritis (OA) of the knee
* OA knee pain present for at least 3 months
* OA knee pain is the predominant (ie, most painful) pain condition
* Patients require medication on at least 4 of 7 days per week to treat OA knee pain for at least 1 month.
* Dissatisfaction with current OA knee pain treatment and willingness to stop taking all pain medications except for the study drug and allowed rescue medication
* Average daily pain rating of at least 5 on a 0 to 10 point numerical rating scale during the 1 week prior to randomization
* Female patients either postmenopausal, surgically sterile or practicing a medically acceptable method of contraception
* Male patients either status post-bilateral vasectomy or using barrier contraception

Exclusion Criteria:

* Knee pain due to a disorder other than OA
* Other pain that can confound the assessment of, or contribute to, pain at the reference knee
* Surgery at the reference knee within 6 months of Screening or a history of joint replacement surgery at the reference knee
* Trauma to the reference knee within 6 months of Screening with active symptoms
* Steroid injections in the reference knee within 3 months of Screening
* Hyaluronic acid injections in the reference knee within 6 months of Screening
* Body Mass Index > 40 kg/m2
* Patient with any protocol-excluded or clinically significant medical, surgical, or medication history that would limit the patient's ability to complete or participate in this clinical trial or could confound the study assessments

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 619 (Actual)
Dates: Start 2012-12-04 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2014-04-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the weekly average of the daily average pain rating | Baseline to end of treatment (Week 15)

SECONDARY OUTCOMES:
Change from baseline in the physical function subscale of the Western Ontario and McMaster University Index of Osteoarthritis Questionnaire (WOMAC) | Baseline to end of treatment (Week 15)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Grünenthal GmbH
Locations (83):
- United States (83):
  - Site 051, Birmingham, Alabama
  - Site 022, Birmingham, Alabama
  - Site 031, Huntsville, Alabama
  - Site 005, Phoenix, Arizona
  - Site 018, Phoenix, Arizona
  - Site 070, Phoenix, Arizona
  - Site 028, Tucson, Arizona
  - Site 081, Chino, California
  - Site 030, El Cajon, California
  - Site 039, Fair Oaks, California
  - Site 061, Fresno, California
  - Site 084, North Hollywood, California
  - Site 080, Roseville, California
  - Site 004, Sacramento, California
  - Site 044, San Diego, California
  - Site 043, Tustin, California
  - Site 010, Walnut Creek, California
  - Site 027, Westlake Village, California
  - Site 011, Bradenton, Florida
  - Site 071, Clearwater, Florida
  - Site 090, Edgewater, Florida
  - Site 060, Jacksonville, Florida
  - Site 015, Jupiter, Florida
  - Site 013, Miami, Florida
  - Site 003, New Port Richey, Florida
  - Site 012, Ocala, Florida
  - Site 032, Orlando, Florida
  - Site 025, Ormond Beach, Florida
  - Site 058, Pembroke Pines, Florida
  - Site 091, Pinellas Park, Florida
  - Site 007, Sarasota, Florida
  - Site 052, Marietta, Georgia
  - Site 033, Perry, Georgia
  - Site 073, Stockbridge, Georgia
  - Site 086, Chicago, Illinois
  - Site 041, Indianapolis, Indiana
  - Site 085, Valparaiso, Indiana
  - Site 088, Towson, Maryland
  - Site 077, Wheaton, Maryland
  - Site 083, New Bedford, Massachusetts
  - Site 021, North Dartmouth, Massachusetts
  - Site 020, Worcester, Massachusetts
  - Site 016, Bingham Farms, Michigan
  - Site 042, Traverse City, Michigan
  - Site 023, St Louis, Missouri
  - Site 087, Grand Island, Nebraska
  - Site 074, Omaha, Nebraska
  - Site 024, Las Vegas, Nevada
  - Site 072, Las Vegas, Nevada
  - Site 009, Albuquerque, New Mexico
  - Site 068, Albany, New York
  - Site 017, Hartsdale, New York
  - Site 056, Greensboro, North Carolina
  - Site 006, High Point, North Carolina
  - Site 078, Wilmington, North Carolina
  - Site 079, Cincinnati, Ohio
  - Site 008, Cincinnati, Ohio
  - Site 069, Cleveland, Ohio
  - Site 001, Columbus, Ohio
  - Site 048, Toledo, Ohio
  - Site 075, Oklahoma City, Oklahoma
  - Site 029, Bend, Oregon
  - Site 067, Medford, Oregon
  - Site 035, Portland, Oregon
  - Site 045, Altoona, Pennsylvania
  - Site 002, Duncansville, Pennsylvania
  - Site 034, Anderson, South Carolina
  - Site 076, Charleston, South Carolina
  - Site 093, Bristol, Tennessee
  - Site 055, Austin, Texas
  - Site 049, Bryan, Texas
  - Site 038, Dallas, Texas
  - Site 089, San Antonio, Texas
  - Site 040, San Antonio, Texas
  - Site 082, Wichita Falls, Texas
  - Site 019, Draper, Utah
  - Site 064, Ogden, Utah
  - Site 059, Salt Lake City, Utah
  - Site 092, Norfolk, Virginia
  - Site 026, Virginia Beach, Virginia
  - Site 066, Bellevue, Washington
  - Site 057, Renton, Washington
  - Site 065, Seattle, Washington